CLINICAL TRIAL: NCT00059397
Title: Hepatitis C: Grading and Staging by MR
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: R03 (DK62765) (completed 2007); R03DK062765 (NIH)
Record Dates: First submitted 2003-04-24; First posted 2003-04-25 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Hepatitis
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis; Hepatitis C

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
To compare MR imaging findings with biopsy for grading and staging early hepatitis C.

ELIGIBILITY:
Referral only

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States